CLINICAL TRIAL: NCT00033865
Title: Yoga as a Treatment for Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sat Bir Singh Khalsa, PhD, Brigham and Women's Hospital, Division of Sleep Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21 AT000066-01A1
Record Dates: First submitted 2002-04-11; First posted 2002-04-12 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia
Keywords: Insomnia; Yoga; Meditation; Behavioral treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Yoga

ARMS (2):
- 1 (Experimental): Yoga treatment for 8 weeks
  Interventions: Behavioral: Yoga, Relaxation Exercises, Sleep Hygiene
- 2 (No Intervention): Sleep hygiene instructions only

INTERVENTIONS:
Behavioral: Yoga, Relaxation Exercises, Sleep Hygiene — Sleep hygiene and relaxation exercises, with additional yoga
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a daily, 8-week treatment for insomnia using yoga, relaxation exercises or sleep hygiene.

DETAILED DESCRIPTION:
Insomnia is a sleep disorder characterized by a chronic difficulty in initiating and maintaining sleep which has a relatively high prevalence and a significant socioeconomic cost. There is good evidence that cognitive and/or physiological arousal, associated with sustained sympathetic activation, is one of the underlying causes of insomnia. Relaxation treatments such as progressive relaxation and meditation which address the cognitive and somatic arousal associated with insomnia have been found to be effective. Yoga is a comprehensive discipline which includes physical exercises, postures, breathing techniques, and meditation, for the purpose of improving health and well being. Research studies have documented the effectiveness of yoga in reducing sympathetic activation and cognitive and somatic arousal and in the treatment of specific medical disorders. Although it has been used and recommended for the treatment of insomnia, its effectiveness has not been evaluated in a randomized, controlled study. The aim of this proposal is to evaluate the effectiveness of yoga, relaxation exercises or sleep hygiene in the treatment of chronic psychophysiological insomnia. A subjective measure of sleep onset latency will be derived from daily sleep diaries, and an objective measure will be drawn from polysomnographic recordings. Sleep onset latency will be evaluated before and after a two month treatment period in a total of 48 young men and women who have been carefully screened for psychiatric and medical disorders. Subjects will be assigned to a yoga, relaxation exercise, or sleep hygiene treatment group. We anticipate that yoga practice will prove to be an effective treatment for insomnia which will yield significant improvements in sleep onset latency. We also anticipate that these improvements will be maintained at long-term follow up evaluation.

ELIGIBILITY:
Inclusion criteria

* A primary complaint of sleep-onset insomnia for at least 6 months.

  * Reside in the metropolitan Boston area

Exclusion Criteria

* No current other nonpharmacological treatment for insomnia.
* Ability or willingness to discontinue use of hypnotic medications.
* No rotating or night shift work, or transcontinental travel throughout the course of the study protocol.
* No recent or anticipated major life stressors over the course of the study protocol (e.g. impending divorce or terminal illness of a relative).

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2001-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sat Bir Singh Khalsa, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital Division of Sleep Medicine, Boston, Massachusetts, United States

REFERENCES:
- [Background] Murtagh DR, Greenwood KM. Identifying effective psychological treatments for insomnia: a meta-analysis. J Consult Clin Psychol. 1995 Feb;63(1):79-89. doi: 10.1037//0022-006x.63.1.79. PMID 7896994
- [Background] Morin CM, Culbert JP, Schwartz SM. Nonpharmacological interventions for insomnia: a meta-analysis of treatment efficacy. Am J Psychiatry. 1994 Aug;151(8):1172-80. doi: 10.1176/ajp.151.8.1172. PMID 8037252
- [Background] Choliz M. A breathing-retraining procedure in treatment of sleep-onset insomnia: theoretical basis and experimental findings. Percept Mot Skills. 1995 Apr;80(2):507-13. doi: 10.2466/pms.1995.80.2.507. PMID 7675582
- [Background] Integration of behavioral and relaxation approaches into the treatment of chronic pain and insomnia. NIH Technology Assessment Panel on Integration of Behavioral and Relaxation Approaches into the Treatment of Chronic Pain and Insomnia. JAMA. 1996 Jul 24-31;276(4):313-8. doi: 10.1001/jama.1996.03540040057033. PMID 8656544
- [Background] Woolfolk RL, Carr-Kaffashan L, McNulty TF. Meditation training as a treatment for insomnia. Behav Ther 1976;7:359-65.
- [Background] Carr-Kaffashan L, Woolfolk RL. Active and placebo effects in treatment of moderate and severe insomnia. J Consult Clin Psychol. 1979 Dec;47(6):1072-80. doi: 10.1037//0022-006x.47.6.1072. No abstract available. PMID 41856
- [Background] Schoicket SL, Bertelson AD, Lacks P. Is sleep hygiene a sufficient treatment for sleep-maintenance insomnia? Behav Ther 1988;19:183-90.
- [Background] Jacobs GD, Rosenberg PA, Friedman R, Matheson J, Peavy GM, Domar AD, Benson H. Multifactor behavioral treatment of chronic sleep-onset insomnia using stimulus control and the relaxation response. A preliminary study. Behav Modif. 1993 Oct;17(4):498-509. doi: 10.1177/01454455930174005. PMID 8216184
- [Background] Koch, U., Volk, S., Heidenreich, T., and Pflug, B. Yoga treatment in psychophysiological insomnia. Journal of Sleep Research 7(Suppl. 2), 137. 1998.
- [Background] Joshi, KS. Yogic treatment of insomnia: An experimental study. Yoga Mimamsa 1992;30:24-26.
- [Derived] Khalsa SBS, Goldstein MR. Treatment of chronic primary sleep onset insomnia with Kundalini yoga: a randomized controlled trial with active sleep hygiene comparison. J Clin Sleep Med. 2021 Sep 1;17(9):1841-1852. doi: 10.5664/jcsm.9320. PMID 33928908